CLINICAL TRIAL: NCT02397590
Title: A Randomized, Open-label, Six-sequence, Three-period, Multiple Dosing Study to Evaluate the Pharmacokinetic Interaction Between Fimasartan and Atorvastatin in Healthy Male Volunteers
Brief Title: Study to Evaluate the Pharmacokinetic Interaction Between Fimasartan and Atorvastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BR-FMS-CT-117
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A Group (Other): Fimasartan (7 days) → wash out (7days) → Atorvastatin (7 days) → wash out (7days) → Fimasartan+Atorvastatin (7 days)
  Interventions: Drug: Fimasartan; Drug: Atorvastatin
- B Group (Other): Fimasartan (7 days) → wash out (7days) → Fimasartan+Atorvastatin (7 days) → wash out (7days) → Atorvastatin (7 days)
  Interventions: Drug: Fimasartan; Drug: Atorvastatin
- C Group (Other): Atorvastatin (7 days) → wash out (7days) → Fimasartan+Atorvastatin (7 days) → wash out (7days) → Fimasartan (7 days)
  Interventions: Drug: Fimasartan; Drug: Atorvastatin
- D Group (Other): Atorvastatin (7 days) → wash out (7days) → Atorvastatin (7 days) → wash out (7days) → Fimasartan+Atorvastatin (7 days)
  Interventions: Drug: Fimasartan; Drug: Atorvastatin
- E Group (Other): Fimasartan+Atorvastatin (7 days) → wash out (7days) → Fimasartan (7 days) → wash out (7days) → Atorvastatin (7 days)
  Interventions: Drug: Fimasartan; Drug: Atorvastatin
- F Group (Other): Fimasartan+Atorvastatin (7 days) → wash out (7days) → Atorvastatin (7 days) → wash out (7days) → Fimasartan (7 days)
  Interventions: Drug: Fimasartan; Drug: Atorvastatin

INTERVENTIONS:
Drug: Fimasartan
Drug: Atorvastatin

SUMMARY:
A phase I clinical trial to compare the pharmacokinetics and safety of fimasartan/Atorvastatin combination tablet and coadministration of fimasartan and Atorvastatin in healthy male volunteers.

DETAILED DESCRIPTION:
After subjects have signed informed consent voluntarily, they go through screening period for within 21 days.

Group 1 period 2 period 3 period A F A F+A B F F+A A C A F+A F D A F F+A E F+A F A F F+A A F

At each period taking Fimasartan, subjects of this Group have blood sampling 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hour after medication(15 times in each period).

At each period taking Atorvastatin, subjects of this Group have blood sampling 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hour after medication(12 times in each period).

At each period taking Fimasartan and Atorvastatin, subjects of this Group have blood sampling 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hour after medication(15 times in each period).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged 19- 50 years at screening.
2. Body weight between 19.0 and 28.0 of ideal body weight (IBW)(kg) = {height (cm) - 100} * 0.9

Exclusion Criteria:

1. History of any illness that may affect the absorption, distribution, metabolism or excretion (hepatobiliary, renal, cardiovascular, endocrine (e.g., hypothyroidism), respiratory, gastrointestinal, hemato-oncology, central nervous system, psychiatric and musculoskeletal system)
2. Hypotension (systolic ≤ 100 mmHg or diastolic ≤ 65 mmHg) or hypertension (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg), measured at screening
3. Evidence of hereditary disease, including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
4. History of gastrointestinal disease (i.g., Crohn's disease, active peptic ulcer) or resection operation that may affect the absorption of the study drug (excluding simple appendectomy or herniorrhaphy)]
5. Participation in any other study within 2 months prior to the first administration of study drug (The finish time of previous study is the day of the last administration of study drug)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
AUC tau,ss | Time Frame: 0~48 hour after medication
Cmax,ss | Time Frame: 0~48 hour after medication

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea